CLINICAL TRIAL: NCT03963492
Title: Intermittent vs. Continuous Walking Training in People With Multiple Sclerosis: a Comparison of Effectiveness
Brief Title: Intermittent vs Continuous Walking in People With Multiple Sclerosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Mount Sinai Rehabilitation Hospital (Other); City University of New York, School of Public Health (Other)
Responsible Party: Principal Investigator, Evan T. Cohen, SHRP Department of Rehabilitation and Movemen, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2019000453
Record Dates: First submitted 2019-05-16; First posted 2019-05-24 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
Keywords: Walking; Gait; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Randomized controlled pre-post study
Who Masked: Outcomes Assessor
Masking Description: Assessors blinded to experimental condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Walking (Active Comparator): Participants in the Continuous Walking (CONT) arm will undergo training 2x/week for 6 weeks for a total plan of 12 training sessions. The intervention for the CONT group will be to complete a 6-minute long walk without rest breaks
  Interventions: Other: Walking
- Interval Walking (Experimental): Participants in the Interval Walking (INT) arm will undergo training 2x/week for 6 weeks for a total plan of 12 training sessions. The intervention for the (INT) group will be to complete three 2-minute-long walks with 2-minute seated rest breaks between each walk
  Interventions: Other: Walking

INTERVENTIONS:
Other: Walking — Participants will undergo training in either the CONT or INT walking interventions 2x/week for 6 weeks for a total plan of 12 training sessions.

SUMMARY:
This study will compare the effectiveness of a traditional, continuous walking rehabilitation program for people with MS to the novel intervention of an intermittent or interval walking rehabilitation program. Half of the participants will receive the continuous walking program while the other half will receive the novel intermittent walking program.

DETAILED DESCRIPTION:
The typical rehabilitation of walking difficulties for people with MS has included practice walking. In general, this includes training to build walking endurance by having the person with MS walk until he/she becomes tired and needs to stop. Although this model has been used successfully to treat people with other diagnoses, it has limited effectiveness in improving walking ability and endurance in people with MS because of fatigue. Recently, a different model has been considered: intermittent or interval walking training. Interval walking training is organized such that seated rest breaks are intentionally interspersed between walking training bouts that end before the person with MS becomes too tired to continue. Exploratory research has shown that people with MS can walk faster and farther when using interval walking training, and may have more improvements in walking ability and endurance after using interval walking training. This study will compare the effectiveness of the traditional model of continuous walking training to the promising new model of interval walking training. This will help to determine whether interval or continuous walking training is superior in improving walking ability and endurance in people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified difficulty walking
* Definitive diagnosis of multiple sclerosis from a neurologist
* Signed an approved consent form
* Ability to ambulate for unaided for 6-minutes continuously with or without an assistive device (e.g. a cane or brace)
* Has not had a multiple sclerosis relapse in the past 6 weeks

Exclusion Criteria:

* Unwilling or unable to complete assessments
* Unwilling or able to complete assessments and or intervention without the use of portable functional electrical stimulation devices
* Medical history of concomitant condition unrelated to multiple sclerosis which may impact results including: other neurological conditions including stroke, Parkinson's disease, or orthopedic, or cardiopulmonary conditions that affect walking
* Had a major change in exercise habits in the past three months
* Individuals reporting change in any disease modifying treatment or steroid use during the past 6 weeks
* Unable to walk for 6 minutes continuously without physical assistance
* Medical history of unstable angina, uncontrolled cardiac dysrhythmias causing symptoms, symptomatic severe aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus or pulmonary infarction, history of deep vein thrombosis, acute myocarditis or pericarditis, acute systemic infection, uncontrolled hypertension, and uncontrolled diabetes
* Has an abnormal response to exercise
* Cannot adhere to protocol
* Determined to be unsafe at the discretion of the research team including individuals unwilling to wear safety "gait belt" during testing or not willing to wear proper footwear.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute Walk Test distance | Baseline, 6 weeks (after intervention), and 12 weeks (6-week follow-up)
  Is a measurement of the distance (in meters) walked at best pace in six minutes.

SECONDARY OUTCOMES:
Change in 12-item Multiple Sclerosis Walking Scale score | Baseline, 6 weeks (after intervention), and 12 weeks (6-week follow-up)
  A survey that measures a participant's perception of how his/her walking ability is affected by multiple sclerosis. The scale ranges from 0-100 with lower scores representing a lesser impact of multiple sclerosis on the participant's walking ability. There are no subscales.
Change in Fatigue Severity Scale score | Baseline, 6 weeks (after intervention), and 12 weeks (6-week follow-up)
  A survey that measures a participant's perception of the impact of the symptom of fatigue on a person's ability to participate in life roles. The scale ranges from from 9-63, with lower scores representing a lower impact of fatigue on the ability to perform the activities listed in the scale.There are no subscales.
Change in Step Length | Baseline, 6 weeks (after intervention), and 12 weeks (6-week follow-up)
  The distance (in centimeters) traversed in one step from initial contact of one foot to the initial contact of the opposite foot.
Change in Step Time | Baseline, 6 weeks (after intervention), and 12 weeks (6-week follow-up)
  The time (in seconds) taken to complete one step from initial contact of one foot to the initial contact of the opposite foot.
Change in Stride Velocity | Baseline, 6 weeks (after intervention), and 12 weeks (6-week follow-up)
  The speed with which it takes a person to complete one stride from initial contact of one foot to the next initial contact of the same foot
Change in Cadence | Baseline, 6 weeks (after intervention), and 12 weeks (6-week follow-up)
  The number of steps (the initial contact of one foot to the initial contact of the opposite foot taken per minute

CONTACTS AND LOCATIONS:
Overall Officials: Evan T Cohen, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Mandell Center for Multiple Sclerosis - Mount Sinai Rehabilitation Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No